CLINICAL TRIAL: NCT02944786
Title: Help Overcoming Pain Early - an Adolescent-centered School Health Prevention Program When Adolescents Have Chronic Pain
Brief Title: Help Overcoming Pain Early - an Adolescent-centered School Health Prevention Program
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205205215
Record Dates: First submitted 2016-10-17; First posted 2016-10-26 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Adolescents; School nurse
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOPE-model (Experimental): Four person-centred health dialogue sessions that include pain/stress management and education about stress and pain.
  Interventions: Behavioral: HOPE-model
- Control (No Intervention): Standard care

INTERVENTIONS:
Behavioral: HOPE-model — There are four sessions of person-centered health dialogues. The sessions also include pain/stress management and education about stress and pain (the HOPE model that is an adolescent-centered school health prevention program when adolescents have chronic pain).
  Arms: HOPE-model

SUMMARY:
The overall aim of the project is to evaluate the Help Overcoming Pain Early model (which includes patient education, person-centered health dialogues and pain/stress management), which is an adolescent-centered school health prevention program when adolescents have chronic pain. This is an intervention that has the hypothesis to support students to manage their chronic pain. The primary outcome is self-efficacy. Secondary outcomes are self-rated health, quality of sleep, pain intensity and school attendance. The project aims to evaluate the intervention through qualitative and quantitative data collection by students and school nurses. The project has a hybrid design, which means that outcomes of the intervention and the evaluation of the implementation are taking place in the same data collection. The results of this project can be of great importance in the early detection of students with chronic pain and promote their confidence in their own ability to manage their symptoms.

DETAILED DESCRIPTION:
School nurses who perform the person-centered health dialogues with the students will have an education, which includes a various of lectures about person-centered health dialogues, stress/pain management and school nurses (over-)generalizations of gender. The project has a hybrid design, which means that outcomes of the intervention and the evaluation of the implementation are taking place in the same data collection.

All students at the participating schools who fulfill the criteria of chronic pain that is mediated by stress, will be invited to participate in the intervention. The participants will be randomized to either group A or group B.

Participants will once report frequency, duration and intensity of pain and they also fill in the questionnaire Center for Epidemiologic Studies Depression Scale for Children.

In the first period of data collection, the group A will get four sessions of person-centered health dialogues. The sessions also include pain/stress management and education about stress and pain (the HOPE model that is an adolescent-centered school health prevention program when adolescents have chronic pain). Group B will be a control group.

All participating school nurses and students will be interviewed about their experiences of the intervention.

In the second period of data collection it will be the other way around, i.e., group B will will get four sessions of person-centered health dialogues. The sessions also include pain/stress management and education about stress and pain (the HOPE model that is an adolescent-centered school health prevention program when adolescents have chronic pain). Group A will be the control group.

All participating school nurses and students will once again be interviewed about their experiences of the intervention.

The primary outcome in the intervention is self-efficacy and this outcome will be measured before and after the intervention in both group A and group B. Secondary outcomes are self-rated health, quality of sleep, pain intensity, and school attendance and these outcomes will also be measured before and after the intervention in both group A and group B.

ELIGIBILITY:
Inclusion Criteria:

* All students who fulfill the criteria of chronic pain that is mediated by stress

Exclusion Criteria:

* Students who cannot speak Swedish or English

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change in Self-Efficacy for Daily Activities (SEDA) score | baseline and 5 weeks after baseline
  Measurement of changes in SEDA from baseline to timepoint 2 that is directly after the intervention period, i.e. week 5 after baseline.
Long term change in Self-Efficacy for Daily Activities (SEDA) score | baseline and 6 months after baseline
  A follow-up measurement of SEDA that will be done at time point 3, i.e. 6 months after baseline.

SECONDARY OUTCOMES:
Change in Minimal Insomnia Symptom Scale (MISS) score | baseline and 5 weeks after baseline
  Measurement of changes in MISS from baseline to timepoint 2 that is directly after the intervention period, i.e. week 5 after baseline.
Long term Change in Minimal Insomnia Symptom Scale (MISS) score | baseline and 6 months after baseline
  A follow-up measurement of MISS that will be done at time point 3, i.e. 6 months after baseline.
Change in Numeric Rating Scale (NRS) for school attendance | baseline and 5 weeks after baseline
  Measurement of changes in NRS school attendance from baseline to timepoint 2 that is directly after the intervention period, i.e. week 5 after baseline.
Long term in Numeric Rating Scale (NRS) of school attendance | baseline and 6 months after baseline
  A follow-up measurement of NRS school attendance that will be done at time point 3, i.e. 6 months after baseline.
Change of Numeric Rating Scale (NRS) score of pain intensity | baseline and 5 weeks after baseline
  Measurement of changes in NRS pain intensity from baseline to timepoint 2 that is directly after the intervention period, i.e. week 5 after baseline.
Long term change in Numeric Rating Scale (NRS) score pain intensity | baseline and 6 months after baseline
  A follow-up measurement of NRS pain intensity that will be done at time point 3, i.e. 6 months after baseline.
Change in Self-Rated Health (SRH) score | baseline and 5 weeks after baseline
  Measurement of changes in SRH from baseline to timepoint 2 that is directly after the intervention period, i.e. week 5 after baseline.
Long term change in Self-Rated Health (SRH) score | baseline and 6 months after baseline
  A follow-up measurement of SRH that will be done at time point 3, i.e. 6 months after baseline.

OTHER OUTCOMES:
Center for Epidemiological Studies Depression Scale for Children (CES-DC) score | Baseline
  A single time point of assessment at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Nilsson, PhD, Principal Investigator — Institute of Health and Care Sciences, University of Gothenburg
Locations (1):
- University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alfven G, Nilsson S. Validity and reliability of a new short verbal rating scale for stress for use in clinical practice. Acta Paediatr. 2014 Apr;103(4):e173-5. doi: 10.1111/apa.12558. Epub 2014 Feb 18. No abstract available. PMID 24533818
- [Result] Barkmann C, Erhart M, Schulte-Markwort M; BELLA Study Group. The German version of the Centre for Epidemiological Studies Depression Scale for Children: psychometric evaluation in a population-based survey of 7 to 17 years old children and adolescents--results of the BELLA study. Eur Child Adolesc Psychiatry. 2008 Dec;17 Suppl 1:116-24. doi: 10.1007/s00787-008-1013-0. PMID 19132311
- [Result] Broman JE, Smedje H, Mallon L, Hetta J. The Minimal Insomnia Symptom Scale (MISS): a brief measure of sleeping difficulties. Ups J Med Sci. 2008;113(2):131-42. doi: 10.3109/2000-1967-221. PMID 18509808
- [Result] Castarlenas E, Sanchez-Rodriguez E, Vega Rde L, Roset R, Miro J. Agreement between verbal and electronic versions of the numerical rating scale (NRS-11) when used to assess pain intensity in adolescents. Clin J Pain. 2015 Mar;31(3):229-34. doi: 10.1097/AJP.0000000000000104. PMID 24699160
- [Result] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Result] Duberg A, Hagberg L, Sunvisson H, Moller M. Influencing self-rated health among adolescent girls with dance intervention: a randomized controlled trial. JAMA Pediatr. 2013 Jan;167(1):27-31. doi: 10.1001/jamapediatrics.2013.421. PMID 23403597
- [Result] Holm S, Ljungman G, Asenlof P, Linton SJ, Soderlund A. Treating youth in pain: Comparing tailored behavioural medicine treatment provided by physical therapists in primary care with physical exercises. Eur J Pain. 2016 Apr;20(4):626-38. doi: 10.1002/ejp.780. Epub 2015 Sep 24. PMID 26399225